CLINICAL TRIAL: NCT07084441
Title: Comparison of Outcomes of Management of Bowel Obstruction
Acronym: COMBO
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, David Flum, Professor and Associate Chair of Research, Director of the Surgical Outcomes Research Center (SORCE), Adjunct Professor, Dept. of Pharmacy, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00020975
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Adhesive Small Bowel Obstruction
Keywords: asbo; sbo; small bowel obstruction; dexamethasone
MeSH Terms: interventions — Dexamethasone; Palliative Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone (Active Comparator): 8 mg IV daily in the morning continued for up to 5 days until SBO is resolved or patient becomes surgical candidate.
  Interventions: Drug: Dexamethasone; Other: Supportive Care
- Supportive Care (Placebo Comparator): Supportive care in both arms includes nasogastric tube (NGT) decompression, hydration, and serial exams to rule out bowel compromise.
  Interventions: Other: Supportive Care

INTERVENTIONS:
Drug: Dexamethasone — *Please see description for dexamethasone + supportive care arm.
  Arms: Dexamethasone
Other: Supportive Care — *Please see description for supportive care arm.

SUMMARY:
The Comparison of Outcomes of Management of Bowel Obstruction (COMBO) trial is a patient-level randomized trial of a short course of dexamethasone + supportive care vs supportive care alone for patients with adhesion-related small bowel obstruction (aSBO). The goal of the COMBO trial is to answer the question: Can Dexamethasone increases the proportion of patients with resolution of aSBO with non-operative management (without complication) based on an established minimal important clinical difference.

DETAILED DESCRIPTION:
Millions of Americans each year experience adhesion-related small bowel obstruction (aSBO), a condition associated with significant morbidity and prolonged hospitalization. Adhesions formed after previous abdominopelvic surgery can cause twisting of the bowel resulting in injury and a cascade of inflammation that results in progressive bowel wall edema with narrowing of the bowel lumen. This leads to or worsens the bowel obstruction. Reversing this inflammation has the potential to reduce the severity and impact of aSBO, hasten the return of bowel function and avoid an emergency operation to treat the obstruction. Dexamethasone, administered intravenously 2-3 times/day for 5-7 days, has been found effective in patients with a form of SBO related to malignancy (malignant ascites or metastatic disease). A Cochrane review evaluated three RCTs of dexamethasone in patients with malignant SBO and found "evidence that dexamethasone…may bring about the resolution of bowel obstruction" and avoid the need for surgical interventionxx . An underappreciated aspect of these RCTs is that almost all patients had a history of abdominopelvic surgery. Since it is difficult to distinguish the extent to which an SBO is caused by adhesions from prior surgery or mass effect related to malignant ascites or metastases, we hypothesize that dexamethasone may be efficacious in resolving aSBO as well.

The Comparison of Outcomes of Management of Bowel Obstruction (COMBO) study is a double-blinded randomized study of a short course of dexamethasone and supportive care vs. supportive care alone for patients with aSBO. The primary outcome is resolution of SBO without operative management and/or major complications as defined using modified National Surgical Quality Improvement Program (NSQIP) criteria. Differences in secondary outcomes-clinical, healthcare utilization and patient-reported outcomes will be explored overall and across subgroups (e.g., based on severity of aSBO, history of aSBO, sex). Reducing inflammation with dexamethasone- a readily available and safe intervention - may improve the likelihood of non-operative management of aSBO and could change the management of millions of patients with this condition.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age recruited from UWMC
* Patients presenting to surgical services through the Emergency Department, diagnosis of SBO, consulted by surgeon, and an urgent or emergency operation is deemed not necessary by surgeon.
* Diagnosis of aSBO is established by;

  1. CT findings consistent with diagnosis of SBO; and
  2. signs and symptoms consistent with SBO; and
  3. Adhesions are the likely cause of SBO (absence of incarcerated hernia, internal hernia, masses, fistula, stricture, volvulus, acute episode of inflammatory bowel disease (IBD) flare, etc.).
* Ability to provide written or electronic informed consent in English and answer teach-back questions

Exclusion Criteria:

* Signs and symptoms of peritonitis with emergency operation planned
* Planned urgent operation within the next 12 hours
* Allergy to dexamethasone
* Surgery within prior 6 weeks
* Unable or unwilling to return or be contacted for and/or complete research surveys
* Currently incarcerated in a detention facility or in police custody (patients wearing a monitoring device can be enrolled) at baseline/screening
* Individuals with latent infections who have an increased risk of infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Resolution of aSBO | 30 days
  The primary outcome is the resolution of aSBO, defined as the absence of obstruction symptoms, in patients receiving dexamethasone + supportive care compared to those receiving supportive care alone

SECONDARY OUTCOMES:
Hospital readmissions - 1 Year | 1 Year
  The outcome for this aim is the comparison of healthcare utilization (e.g., readmissions) between the dexamethasone and supportive care groups
Patient-Reported Outcomes (PROs) - GIQLI | 30 days
  The outcome will be the comparison of patient-reported outcomes of gastrointestinal quality of life (GIQLI) between the dexamethasone and supportive care groups.
Hospital readmissions - 30 day | 30 day
  The outcome for this aim is the comparison of healthcare utilization (e.g., readmissions) between the dexamethasone and supportive care groups

CONTACTS AND LOCATIONS:
Overall Officials: David Flum, MD, Principal Investigator — University of Washington

IPD SHARING:
Plan to Share IPD: No